CLINICAL TRIAL: NCT03026491
Title: Chewing Function in Children With Repaired Esophageal Atresia-tracheoesophageal Fistula
Brief Title: Chewing in Children With Repaired Esophageal Atresia-tracheoesophageal Fistula
Status: Completed | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, SELEN SEREL ARSLAN, Principal Investigator, Hacettepe University
Other Study IDs: EA-TEF
Record Dates: First submitted 2017-01-15; First posted 2017-01-20 (Estimated); Last update posted 2017-08-09 (Actual); Status verified 2017-08

CONDITIONS: Chewing Problem

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Children with chewing dysfunction: Descriptive characteristics including age, height, weight, transition time to additional food, meal time, number of meals, initial teething time, and number of teeth, were noted. The presence of open mouth, open bite, high palate, gag reflex, and oral hygiene were scored as absent or present as an observational oral motor assessment. Chewing evaluation was performed and scored with the Karaduman Chewing Performance Scale (KCPS). The International Dysphagia Diet Standardisation Initiative (IDDSI) was used to determine the tolerated food texture of children.
  Interventions: Other: Chewing evaluation
- Children without chewing dysfunction: Descriptive characteristics including age, height, weight, transition time to additional food, meal time, number of meals, initial teething time, and number of teeth, were noted. The presence of open mouth, open bite, high palate, gag reflex, and oral hygiene were scored as absent or present as an observational oral motor assessment. Chewing evaluation was performed and scored with the Karaduman Chewing Performance Scale (KCPS). The International Dysphagia Diet Standardisation Initiative (IDDSI) was used to determine the tolerated food texture of children.
  Interventions: Other: Chewing evaluation

INTERVENTIONS:
Other: Chewing evaluation — Each child was required to bite and chew a standardized biscuit while chewing video recording. Chewing function was scored with the Karaduman Chewing Performance Scale (KCPS).

SUMMARY:
The investigators aim to evaluate chewing function in children with repaired esophageal atresia-tracheoesophageal fistula (EA-TEF). Patients with repaired EA-TEF will be evaluated for age, sex, type of atresia. Each child will be required to bite and chew a standardized biscuit. Chewing function will be scored with the Karaduman Chewing Performance Scale (KCPS). The International Dysphagia Diet Standardisation Initiative (IDDSI) will be used to determine the tolerated food texture of children.

DETAILED DESCRIPTION:
The diet of children with normal feeding skills includes a combination of liquid, semisolid and/or solid foods. Chewing dysfunction (CD) in children may cause restrictions in solid food intake, thereby may result in insufficient food intake and delay in growth. It is aim to evaluate chewing function in children with repaired esophageal atresia-tracheoesophageal fistula (EA-TEF). Patients with repaired EA-TEF will be evaluated for age, sex, type of atresia. Each child will be required to bite and chew a standardized biscuit. Chewing function will be scored with the Karaduman Chewing Performance Scale (KCPS). The International Dysphagia Diet Standardisation Initiative (IDDSI) will be used to determine the tolerated food texture of children.

ELIGIBILITY:
Inclusion Criteria:

* Children with repaired esophageal atresia-tracheoesophageal fistula, without airway aspiration, intact airway closure

Exclusion Criteria:

* Children without repaired esophageal atresia-tracheoesophageal fistula, with airway aspiration, insufficient airway closure

Ages: 24 Months to 192 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children with repaired esophageal atresia-tracheoesophageal fistula
Sampling Method: Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2017-03-01 (Actual); Study Completion 2017-04-01 (Actual)

PRIMARY OUTCOMES:
Chewing function will be scored with the Karaduman Chewing Performance Scale (KCPS) | 10 minutes
  Chewing function will be evaluated

SECONDARY OUTCOMES:
Observational oral motor assessment will be performed | 15 minutes
  The presence of open mouth posture, open bite, tongue thrust, high palate will be noted as ''absent'' or ''present''. The body position, hyper/hyposensitivity, jaw, lips/cheeks and tongue movements of the children will be assessed .

CONTACTS AND LOCATIONS:
Overall Officials: SELEN SEREL ARSLAN, PhD, Principal Investigator — Hacettepe University

IPD SHARING:
Plan to Share IPD: No